CLINICAL TRIAL: NCT04537923
Title: A Randomized, Phase 3, Open-label Trial Comparing the Effect of the Addition of Tirzepatide Once Weekly Versus Insulin Lispro (U100) Three Times Daily in Participants With Type 2 Diabetes Inadequately Controlled on Insulin Glargine (U100) With or Without Metformin (SURPASS-6)
Brief Title: A Study of Tirzepatide (LY3298176) Versus Insulin Lispro (U100) in Participants With Type 2 Diabetes Inadequately Controlled on Insulin Glargine (U100) With or Without Metformin
Acronym: SURPASS-6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17204; I8F-MC-GPHD (Other: Eli Lilly and Company); 2020-000284-23 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-09-03 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes
Keywords: glucose-dependent insulinotropic polypeptide (GIP); glucagon-like peptide-1 (GLP-1); GIP/GLP-1 dual receptor agonist; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- Insulin Lispro (Active Comparator): Insulin lispro 100 units per milliliter (U100) administered SC three times a day.
  Interventions: Drug: Insulin Lispro (U100)

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Insulin Lispro (U100) — Administered SC
  Other Names: LY275585
  Arms: Insulin Lispro

SUMMARY:
The purpose of this study is to compare the safety and efficacy of the study drug tirzepatide to insulin lispro (U100) three times a day in participants with type 2 diabetes that are already on insulin glargine (U100), with or without metformin.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus (T2DM)
* Have HbA1c between ≥7.5% and ≤11%
* Have been treated for at least 90 days prior to day of screening with once or twice daily basal insulin with or without stable dose of metformin ≥1500 mg/day and up to maximum approved dose per country specific approved label, sulfonylureas or dipeptidyl peptidase 4 inhibitors
* Be of stable weight (± 5%) for at least 90 days
* Have a BMI ≥23 kilograms per meter squared (kg/m²) and ≤45 kg/m² at screening

Exclusion Criteria

* Have type 1 diabetes mellitus
* Have had chronic or acute pancreatitis any time prior to study entry
* Have proliferative diabetic retinopathy or diabetic macular edema or nonproliferative diabetic retinopathy requiring immediate or urgent treatment
* Have disorders associated with slowed emptying of the stomach, have had any stomach surgeries for the purpose of weight loss, or are chronically taking drugs that directly affect gastrointestinal motility
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months
* Have an estimated glomerular filtration rate <30 mL/minute/1.73 m² [for participants on metformin, estimated glomerular filtration rate <45 mL/min/1.73 m2 (or lower than the country-specific threshold for using the protocol-required dose of metformin per local label)]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (135):
- United States (40):
  - Syed Research Consultants Llc, Sheffield, Alabama
  - Valley Research, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Huntington Park, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - National Research Institute - Huntington Park, Panorama City, California
  - National Research Institute (NRI) - Santa Ana, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - University of Colorado, Aurora, Colorado
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - I R & Health Center, Inc., Hialeah, Florida
  - Sun Coast Clinical Research, Inc, New Port Richey, Florida
  - South Broward Research, Pembroke Pines, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - J H. Stroger Hosp of Cook Co, Chicago, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Capital Diabetes and Endocrine Associates, Camp Springs, Maryland
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Glacier View Research Institute - Endocrinology, Kalispell, Montana
  - Southern Nh Diabetes and Endocrinology, Nashua, New Hampshire
  - Albany Medical College, Albany, New York
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Intend Research, LLC, Norman, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Dallas Diabetes Research Center, Dallas, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - North Hills Medical Research, North Richland Hills, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (12):
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Investigaciones Medicas Imoba Srl, CABA, Buenos Aires
  - Instituto Centenario, CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Rosario (IIC-Rosario)- Sanatorio Delta, Rosario, Buenos Aires
  - CIPADI, Godoy Cruz, Mendoza Province
  - Instituto Médico Catamarca, Rosario, Santa Fe Province
  - Instituto Médico Especializado (IME), Buenos Aires
  - Asociación de Beneficencia Hospital Sirio Libanés, Buenos Aires
  - CENUDIAB, Ciudad Autónoma de Buenos Aire
  - Centro Diabetologico Dr Waitman, Córdoba
  - Centro Medico Privado San Vicente Diabetes, Córdoba
  - Sanatorio Parque, Salta
- AZ Damiaan Oostende, Ostend, Belgium
- Brazil (15):
  - Centro de Pesq. em Diabetes e Doencas Endocrino Metabol., Fortaleza, Ceará
  - CEDOES, Vitória, Espírito Santo
  - Cline Research Center, Curitiba, Paraná
  - QUANTA - Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Centro de Pesquisas em Diabetes, Porto Alegre, Rio Grande do Sul
  - Hospital PUC-CAMPINAS, Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos EPP Ltda, São Bernardo do Campo, São Paulo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - CPCLIN, São Paulo, São Paulo
  - Instituto Brasil de Pesquisa Clínica - IBPCLIN, Rio de Janeiro
  - IPEC - Instituto de Pesquisa Clínica, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - BR Trials - Ensaios Clínicos e Consultoria Ltda, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Czechia (4):
  - Diabetologicka ordinace pro dospele, Krnov, Moravskoslezský kraj
  - Diabetologicka a obezitologicka ambulance, České Budějovice
  - Diahelp s.r.o., Interni a diabetologicka ambulance, Pardubice
  - ResTrial s.r.o., Prague
- Germany (9):
  - Schwerpunktpraxis für Diabetes, Hof, Bavaria
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Medizentrum Essen-Borbeck, Essen, North Rhine-Westphalia
  - Zentrum für klinische Studien, Saint Ingbert, Saarland
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - MVZ im Altstadt-Carree Fulda GmbH, Fulda
  - Diabetologische Schwerpunktpraxis Harburg, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
  - Gemeinschaftspraxis Dr. med. Josef und Wilma Großkopf, Wallerfing
- Greece (4):
  - Iatriko Palaiou Falirou, Medical Center, Palaió Fáliro, Athens
  - Athens Euroclinic, Athens, Attica
  - General Hospital of Thessaloniki Papageorgiou, N. Efkarpia, Thessaloniki
  - Thermi Clinic, Thermi, Thessaloniki
- Hungary (4):
  - Belinus Bt, Debrecen, Hajdú-Bihar
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Intezet, Debrecen, Hajdú-Bihar
  - Szent Margit Rendelőintézet Nonprofit Kft, Budapest
  - TRANTOR'99 Bt. Anyagcsere Centrum, Budapest
- Italy (4):
  - Policlinico Mater Domini, Germaneto, Catanzaro
  - Casa di Cura Multimedica-Policlinico Multispecialistico, Sesto San Giovanni, MI
  - Ospedale Luigi Sacco, Milan
  - Policlinico Univ. Agostino Gemelli, Roma
- Mexico (5):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesida, Guadalajara, Jalisco
  - Unidad de patologia Clinica, Guadalajara, Jalisco
  - Centro de Inv. Medica de Occidente, SC, Zapopan, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, N.L.
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Madero, Tamaulipas
- Puerto Rico (2):
  - Centro de Endocrinologia y Nutricion del Turabo, Caguas, PR
  - Paola Mansilla-Letelier, MD, Guaynabo, PR
- Romania (12):
  - SC Endodigest SRL, Oradea, Bihor County
  - S. C. Grandmed S.R.L., Oradea, Bihor County
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - SC Gama Diamed SRL, Mangalia, Constanța County
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - SC Cosamext SRL, Târgu Mureş, Mureș County
  - SC Diabmed Dr Popescu Alexandrina SRL, Ploieşti, Prahova
  - SC Dianutrilife Medica SRL, Ploieşti, Prahova
  - Centrul Medical Dr. Negrisanu, Timișoara, Timiș County
  - Cabinetul Medical Nicodiab SRL, Bucharest
  - SC Nutrilife SRL, Bucharest
  - Milena Sante SRL, Galati
- Russia (8):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Scientific and Clinical Center for Precision and Regenerative Medicine, Kazan'
  - Pirogov Russian National Research Medical University, Moscow
  - First Moscow State Medical University, Moscow
  - City Consultative and Diagnostic Center #1, Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of Healthcare Institution, Saint Petersburg
  - St.Petersburg Polyclinic #117, Saint Petersburg
  - SPb GUZ "Diagnostic Center #85", Saint Petersburg
- Slovakia (5):
  - Diacrin s.r.o., Bratislava, Bratislava Region
  - MediVet s.r.o., Malacky, Bratislava Region
  - Human care s.r.o., Košice, Slovak Republic
  - Diabetes care s.r.o., Hnúšťa
  - Areteus s.r.o., Trebišov
- Spain (5):
  - Hospital Quiron Infanta Luisa, Seville, Andalusia
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario De Ferrol - Hospital Naval, Ferrol, La Coruna
  - Clínica Juaneda, Palma de Mallorca
  - Hospital Universitario Virgen Macarena, Seville
- Turkey (Türkiye) (5):
  - Baskent Universitesi Adana Uygulama ve Arastirma Merkezi Yuregir Hastanesi, Adana
  - Akdeniz University Medical Faculty, Antalya
  - Aydin Adnan Menderes Universitesi, Aydin
  - Gaziantep University Medical Faculty, Gaziantep
  - Inonu Universitesi, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Rosenstock J, Frias JP, Rodbard HW, Tofe S, Sears E, Huh R, Fernandez Lando L, Patel H. Tirzepatide vs Insulin Lispro Added to Basal Insulin in Type 2 Diabetes: The SURPASS-6 Randomized Clinical Trial. JAMA. 2023 Nov 7;330(17):1631-1640. doi: 10.1001/jama.2023.20294. PMID 37786396
- See also: A Study of Tirzepatide (LY3298176) Versus Insulin Lispro (U100) in Participants With Type 2 Diabetes Inadequately Controlled on Insulin Glargine (U100) With or Without Metformin (SURPASS-6) — https://trials.lillytrialguide.com/en-US/trial/11LK1nZPXq4bEVBd2Mdi2i

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 mg Tirzepatide: Participants received 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
- 10 mg Tirzepatide: Participants received 10 mg tirzepatide administered SC once a week .
- 15 mg Tirzepatide: Participants received 15 mg tirzepatide administered SC once a week.
- Insulin Lispro: Participants received Insulin lispro 100 units per milliliter (U100) administered SC three times a day.
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Started | 243 | 238 | 236 | 711
Received at Least One Dose of Study Drug | 243 | 238 | 236 | 708
Completed | 228 | 228 | 225 | 623
Not Completed | 15 | 10 | 11 | 88
Not completed — Adverse Event | 2 | 1 | 2 | 4
Not completed — Death | 3 | 3 | 1 | 11
Not completed — Lost to Follow-up | 1 | 2 | 1 | 6
Not completed — Physician Decision | 1 | 0 | 2 | 5
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 4 | 58
Not completed — Missed study visits | 2 | 0 | 0 | 3
Not completed — Sponsor's decision | 0 | 0 | 1 | 1
Not completed — Safety reasons | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 5 mg Tirzepatide: Participants received 5 mg tirzepatide administered SC once a week.
- 10 mg Tirzepatide: Participants received 10 mg tirzepatide administered SC once a week.
- Insulin Lispro: Participants received Insulin lispro (U100) administered SC three times a day.
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro | Total
Number analyzed (Participants) | 243 | 238 | 236 | 711 | 1428
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.00 (10.18) | 59.60 (9.41) | 58.20 (9.62) | 59.00 (9.74) | 58.80 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 149 | 133 | 398 | 824
  Male | 99 | 89 | 103 | 313 | 604
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 148 | 142 | 149 | 446 | 885
  Not Hispanic or Latino | 95 | 93 | 87 | 261 | 536
  Unknown or Not Reported | 0 | 3 | 0 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 2 | 3
  Asian | 2 | 0 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 9 | 11 | 26 | 57
  White | 230 | 224 | 220 | 671 | 1345
  More than one race | 0 | 5 | 2 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 70 | 70 | 70 | 207 | 417
  Belgium | 0 | 1 | 0 | 1 | 2
  Brazil | 47 | 47 | 46 | 141 | 281
  Czechia | 10 | 9 | 9 | 29 | 57
  Germany | 7 | 8 | 8 | 24 | 47
  Greece | 2 | 2 | 2 | 9 | 15
  Hungary | 4 | 4 | 2 | 9 | 19
  Italy | 1 | 2 | 1 | 2 | 6
  Mexico | 19 | 20 | 20 | 59 | 118
  Romania | 14 | 14 | 12 | 38 | 78
  Russia | 19 | 17 | 19 | 52 | 107
  Slovakia | 16 | 13 | 15 | 39 | 83
  Spain | 5 | 3 | 3 | 14 | 25
  Turkey | 1 | 0 | 1 | 2 | 4
  United States | 28 | 28 | 28 | 85 | 169
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.89 (0.97) | 8.78 (0.98) | 8.74 (1.01) | 8.81 (0.96) | 8.80 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (Pooled Doses of Tirzepatide 5 mg, 10 mg and 15 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomly assigned participants who took at least 1 dose of study drug and had a baseline and at least 1 post-baseline value for this analysis, excluding participants discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug. This analysis was planned to measure the outcome for pooled 5 mg, 10 mg and 15 mg tirzepatide.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Groups:
- Pooled 5 mg/10 mg/15 mg Tirzepatide: Participants received either 5 mg or 10 mg or 15 mg tirzepatide administered SC once a week.
Arm/Group | Pooled 5 mg/10 mg/15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 708 | 692
Percentage of HbA1c | -2.26 (0.048) | -1.16 (0.049)
Statistical Analysis 1: Comparison: Pooled 5 mg/10 mg/15 mg Tirzepatide vs Insulin Lispro; Test type: Non-Inferiority — 0.3% noninferiority margin; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.10, 95% CI 2-sided [-1.24 to -0.97]

2. Secondary Outcome: Change From Baseline in HbA1c
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. LS mean was determined by MMRM model with covariates Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomly assigned participants who took at least 1 dose of study drug and had a baseline and at least 1 post-baseline value for this analysis, excluding participants discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 241 | 234 | 233 | 692
Percentage of HbA1c | -2.05 (0.082) | -2.27 (0.083) | -2.46 (0.084) | -1.16 (0.049)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Non-Inferiority — 0.3% noninferiority margin; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.89, 95% CI 2-sided [-1.08 to -0.70]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Non-Inferiority — 0.3% noninferiority margin; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.11, 95% CI 2-sided [-1.30 to -0.92]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Non-Inferiority — 0.3% noninferiority margin; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.30, 95% CI 2-sided [-1.49 to -1.11]

3. Secondary Outcome: Percentage of Participants With HbA1c Target Values <7.0%
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 242 | 238 | 236 | 708
Percentage of participants | 61.04 | 75.64 | 79.86 | 36.69
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 3.13, 95% CI 2-sided [2.25 to 4.36]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.16, 95% CI 2-sided [4.27 to 8.88]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 7.94, 95% CI 2-sided [5.37 to 11.75]

4. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model with Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 241 | 234 | 233 | 694
Kilograms (kg) | -6.9 (0.37) | -9.9 (0.37) | -12.0 (0.38) | 3.8 (0.22)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -10.7, 95% CI 2-sided [-11.5 to -9.9]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.7, 95% CI 2-sided [-14.5 to -12.9]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -15.9, 95% CI 2-sided [-16.7 to -15.0]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: LS mean was determined by MMRM model with variables Baseline + Pooled Country + Baseline metformin Use (Yes, No) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 241 | 235 | 233 | 694
milligram per Deciliter (mg/dL) | -33.2 (3.28) | -43.0 (3.32) | -41.6 (3.42) | -10.0 (1.99)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -23.2, 95% CI 2-sided [-30.8 to -15.7]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -33.0, 95% CI 2-sided [-40.6 to -25.4]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -31.6, 95% CI 2-sided [-39.3 to -23.8]

6. Secondary Outcome: Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Post meal, Midday Premeal, Midday 2-hour Post meal, Evening Premeal, Evening 2-hour Post meal and Bedtime. The daily average was calculated as the average of the 7 blood glucose values collected on a particular day. LS mean was determined by MMRM model with variables Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL/day
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 219 | 210 | 204 | 574
mg/dL/day | -56.7 (1.80) | -61.5 (1.85) | 67.6 (1.86) | -55.8 (1.13)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p = 0.682, Mixed Models Analysis; LS Mean Difference = -0.9, 95% CI 2-sided [-5.0 to 3.3]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p = 0.010, Mixed Models Analysis; LS Mean Difference = -5.6, 95% CI 2-sided [-9.9 to -1.4]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -11.8, 95% CI 2-sided [-16.0 to -7.5]

7. Secondary Outcome: Percentage of Participants Who Achieved HbA1c Target Value of <7.0% Without Hypoglycemia
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 241 | 234 | 233 | 692
Percentage of participants | 52.70 | 70.05 | 75.12 | 13.41
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.19, 95% CI 2-sided [5.66 to 11.83]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 16.90, 95% CI 2-sided [11.44 to 24.96]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 21.85, 95% CI 2-sided [14.49 to 32.93]

8. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5% is reported here.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 242 | 238 | 236 | 708
Percentage of participants | 64.19 | 79.21 | 83.15 | 6.34
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.25, 95% CI 2-sided [18.36 to 43.46]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 58.90, 95% CI 2-sided [36.76 to 94.39]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 77.76, 95% CI 2-sided [47.49 to 127.33]

9. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and two overall summary scores: physical component summary (PCS) and mental component summary (MCS) scores. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. PCS score is reported here. PCS domain is scored by summing individual items and transforming scores into a 0 to 100 scale with higher scores indicating better health status or functioning. LS mean was determined by analysis of covariance (ANCOVA) model with variables Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 222 | 217 | 199 | 599
score on a scale | 1.0 (0.46) | 1.7 (0.46) | 1.7 (0.48) | -0.6 (0.28)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p = 0.005, ANCOVA; LS Mean Difference = 1.5, 95% CI 2-sided [0.5 to 2.6]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 2.3, 95% CI 2-sided [1.2 to 3.3]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 2.2, 95% CI 2-sided [1.2 to 3.3]

10. Secondary Outcome: Change From Baseline in 36-Item SF-36 Mental Component Summary (MCS) Score
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and two overall summary scores: physical component summary (PCS) and mental component summary (MCS) scores. MCS consisted of social functioning, vitality, mental health, and role-emotional scales. MCS score is reported here. MCS domain is scored by summing individual items and transforming scores into a 0 to 100 scale with higher scores indicating better health status or functioning. LS mean was determined by ANCOVA model with variables Baseline + Pooled Country + Baseline Metformin Use (Yes, No) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
Number analyzed (Participants) | 222 | 217 | 199 | 599
score on a scale | 0.3 (0.59) | 1.5 (0.59) | 0.7 (0.62) | -1.3 (0.36)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p = 0.020, ANCOVA; LS Mean Difference = 1.6, 95% CI 2-sided [0.3 to 2.9]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 2.8, 95% CI 2-sided [1.5 to 4.2]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Lispro; Test type: Superiority; p = 0.004, ANCOVA; LS Mean Difference = 2.1, 95% CI 2-sided [0.7 to 3.5]

ADVERSE EVENTS:
Time Frame: Baseline up to week 56
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Lispro
All-Cause Mortality (participants affected / at risk) | 3/243 | 3/238 | 1/236 | 11/708
Serious Adverse Events (participants affected / at risk) | 20/243 | 16/238 | 17/236 | 81/708
Other Adverse Events (participants affected / at risk) | 94/243 | 116/238 | 121/236 | 99/708
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=243) | 10 mg Tirzepatide (N=238) | 15 mg Tirzepatide (N=236) | Insulin Lispro (N=708)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bullous erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Covid-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 7 (7)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oophoritis (Infections and infestations) | 0/144 (0) | 0/149 (0) | 0/133 (0) | 1/396 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (18) | 1 (1) | 28 (84)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/144 (0) | 0/149 (0) | 0/133 (0) | 1/396 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/144 (1) | 0/149 (0) | 0/133 (0) | 0/396 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthrodesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal cryoablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=243) | 10 mg Tirzepatide (N=238) | 15 mg Tirzepatide (N=236) | Insulin Lispro (N=708)
Constipation (Gastrointestinal disorders) | 6 (9) | 8 (8) | 14 (19) | 4 (9)
Diarrhoea (Gastrointestinal disorders) | 29 (46) | 36 (66) | 26 (49) | 17 (22)
Dyspepsia (Gastrointestinal disorders) | 15 (16) | 27 (47) | 27 (34) | 4 (4)
Nausea (Gastrointestinal disorders) | 33 (71) | 49 (80) | 61 (161) | 8 (11)
Vomiting (Gastrointestinal disorders) | 11 (14) | 21 (35) | 30 (80) | 4 (4)
Covid-19 (Infections and infestations) | 28 (28) | 19 (19) | 21 (23) | 72 (73)
Decreased appetite (Metabolism and nutrition disorders) | 20 (81) | 28 (84) | 40 (128) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT04537923/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT04537923/SAP_001.pdf